CLINICAL TRIAL: NCT03133416
Title: Platelet-rich Plasma Injections and Physiotherapy in the Treatment of Chronic Rotator Cuff Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20160105R; MOST 105-2314-B-341-003 - (Other Grant/Funding Number: Ministry of Science and Technology); MOST 106-2314-B-341-006 - (Other Grant/Funding Number: Ministry of Science and Technology)
Record Dates: First submitted 2017-04-12; First posted 2017-04-28 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-01

CONDITIONS: PRP Injection Only; Physiotherapy Only; PRP and Physiotherapy
Keywords: rotator cuff tendinopathy; rotator cuff tear; platelet-rich plasma; physiotherapy; exercise
MeSH Terms: conditions — Rotator Cuff Injuries; Motor Activity | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRP preparation (Active Comparator): PRP will be prepared by taking 10ml venous blood which is then mixed with 2ml of thrombin and centrifuged in a specially designed tube at 3400 rotations per minute (rpm) for 15 minutes. Then about 2ml PRP will be extracted, and will be infiltrated to the lesion site under ultrasound guidance. The injection technique is similar to that described by Kesikburun .21 Patients in group 1 or group 3 will receive 2 injections of PRP, with 1 month interval.
  Interventions: Other: PRP preparation
- Physiotherapy (Active Comparator): Physiotherapy includes hot pack, electric therapy and therapeutic exercise, which will be supervised by a senior physical therapist. The therapeutic exercise consists of active and passive stretch, and strengthening exercise of the rotator cuff, the shoulder girdle, and the pectoral muscles, 3 times a week, and will continue for 1.5 months. After 1.5 months' supervised training, home program exercise follows and will be continued for another 1.5 months.
  Interventions: Device: Physiotherapy
- PRP and physiotherapy (Active Comparator): PRP will be prepared by taking 10ml venous blood which is then mixed with 2ml of thrombin and centrifuged in a specially designed tube at 3400 rotations per minute (rpm) for 15 minutes. Then about 2ml PRP will be extracted, and will be infiltrated to the lesion site under ultrasound guidance. The injection technique is similar to that described by Kesikburun .21 Patients in group 1 or group 3 will receive 2 injections of PRP, with 1 month interval;Physiotherapy includes hot pack, electric therapy and therapeutic exercise, which will be supervised by a senior physical therapist. The therapeutic exercise consists of active and passive stretch, and strengthening exercise of the rotator cuff, the shoulder girdle, and the pectoral muscles, 3 times a week, and will continue for 1.5 months. After 1.5 months' supervised training, home program exercise follows and will be continued for another 1.5 months.
  Interventions: Other: PRP and physiotherapy

INTERVENTIONS:
Other: PRP preparation
  Arms: PRP preparation
Device: Physiotherapy
  Arms: Physiotherapy
Other: PRP and physiotherapy
  Arms: PRP and physiotherapy

SUMMARY:
The investigators aim to investigate whether combination of PRP injection with physiotherapy program could produce superior effect than either treatment alone.

DETAILED DESCRIPTION:
Rotator cuff (RC) tears are a common source of shoulder pain and account for more than 4.5 million physician visits per year. In the overall population, the prevalence of RC tear is 20.7% and rises to 50% among patients older than 80 years. Partial-thickness and full-thickness RC tears has also been reported in 30% to 50% of the population aged older than 50 years. RC tears cause shoulder dysfunction, interfere daily activity, and may reduce quality of life. Treatment of RC tear includes surgical and conservative treatment. Considering operative risk, high possibility of re-tear after operation, and possible tendon healing with non-surgical treatment, for patients with a partial-thickness tear or a small full-thickness tear, conservative treatment is usually tried first. Previous report found that conservative treatment might be effective in 73% to 80% of cases with full-thickness tear of the rotator cuff. Conservative treatment of RC tear consists of rest, physiotherapy (including therapeutic exercise), non-steroidal anti-inflammatory drugs, and corticosteroid or hyaluronate subacromial injections. A. In addition, exercise has also been proven effective in the management of RC tear. In spite of the advanced surgical techniques and conservative methods, healing of RC tear remains problematic due to poor vascularization at the lesion site and failure to restore normal enthesis (tendon-bone junction) histology. Over past few years platelet-rich plasma (PRP) presents an attractive option to improve and accelerate healing of the rotator cuff lesion. PRP is defined as a portion of the plasma fraction of autologous blood having a platelet concentration above baseline (usually 2X to 4X). It is derived from centrifuging whole blood, and contains numerous growth factors, including platelet-derived growth factor, vascular endothelial growth factor, transforming growth factor, fibroblast growth factor, epidermal growth factor, hepatocyte growth factor, and insulin-like growth factor. Because of the increased concentration and release of growth factors, PRP can potentially enhance the recruitment and proliferation of tenocytes, stem cells, and endothelial cells. Given the autologous nature of PRP, safety concerns are minimal. Relative contraindications include patients with a history of thrombocytopenia, use of anticoagulants, tumor, metastatic disease, active infection, or pregnancy. Up to now no documented cases of carcinogenesis or tumor growth associated with the use of PRP has been reported. Previous studies showed using autologous leukocyte- and platelet-rich fibrin could increase vascularization during early healing of chronic rotator cuff tear, and that ultrasound-guided PRP injection is superior to dry needling in patients with supraspinatus tendon lesion. However, in a 1-yr randomized controlled trial with combination of 6 week physiotherapy program, PRP injection did not produce extra effect than placebo injection. Because controversy exists with regard to the effect of PRP injection, the investigators aim to investigate whether combination of PRP injection with physiotherapy program could produce superior effect than either treatment alone.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic rotator cuff tendinopathy, including small (<1cm) rotator cuff tear (partial or full-thickness), proven by ultrasound.
2. Duration of symptom longer than 1 month.
3. Aged ≥20 years old.

Exclusion Criteria:

1. Fracture, dislocation, or arthritis of the shoulder,
2. Previous shoulder joint surgery,
3. Rotator cuff tear with size ≥ 1cm,
4. Calcification of rotator cuff tendons,
5. Severe medical comorbidities, e.g., malignant neoplasms, blood dyscrasia, and serious infection, etc.,
6. Pregnancy,
7. Cognitive impairment (Mini-Mental Status Examination < 24),
8. Hypersensitive to thrombin.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Change of the VAS for pain | Clinical evaluation will be conducted at pre-treatment, post-treatment 1.5 months and post-treatment 3 months and post-treatment 6 months after treatments.
  The VAS pain scores during Neer test will be obtained using a horizontal lines of 100 mm, with 0 on the left indicating no pain and 100 on the right indicating very severe pain. A VAS has been shown to be reliable and sensitive for quantifying pain, with test-retest reliability of >0.90.28 In previous studies of patients treated for various shoulder disorders, the responsiveness of VAS for pain was moderate to good.

SECONDARY OUTCOMES:
the active ROM | Clinical evaluation will be conducted at pre-treatment, post-treatment 1.5 months and post-treatment 3 months and post-treatment 6 months after treatments.
  The maximal active ROMs of the affected shoulder will be measured using a goniometer under the guidelines of the American Academy of Orthopedic Surgeons. These measurements included abduction in the frontal plane, forward flexion, internal rotation, and external rotation with the arm at 0 degrees of abduction.
SPADI | Clinical evaluation will be conducted at pre-treatment, post-treatment 1.5 months and post-treatment 3 months and post-treatment 6 months after treatments.
  The SPADI is a self-administered questionnaire to assess the pain and disability associated with shoulder diseases. It consists of 13 items being divided into 2 subclasses, 5 items for pain and 8 items for disabilities. The total SPADI score, which ranges between 0 and 100, is calculated by averaging the scores from the pain and disabilities subclasses.
SF-36 | Clinical evaluation will be conducted at pre-treatment, post-treatment 1.5 months and post-treatment 3 months and post-treatment 6 months after treatments.
  The SF-36 is a 36-item questionnaire that evaluates the quality of life . It is composed of eight subscales: physical functioning, physical role, bodily pain, general health, vitality, social functioning, emotional role, and mental health. Each subscale has a score range of 0-100, with a higher score indicating better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Lin-Fen Hsieh, M.D, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- ShinKongHospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided